CLINICAL TRIAL: NCT03460626
Title: Evaluation of Aromatherapy on Academic Stress: A Randomized Placebo Controlled Clinical Trial
Brief Title: Evaluation of Aromatherapy on Academic Stress
Acronym: (EAS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Atta Abbas Naqvi, Co-Investigator, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IAU-ATCT
Record Dates: First submitted 2018-02-19; First posted 2018-03-09 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Stress; Academic Underachievement Disorder
Keywords: stress; pharmacy students; Saudi Arabia
MeSH Terms: interventions — lavender oil

STUDY DESIGN:
Intervention Model Description: The students will be divided into three groups randomly as Group-I (Control group: treated with a placebo that is an odorless oil without any therapeutic effect), Group-II (Treated group: administered with lavender oil) and Group-III (Untreated group)
Who Masked: Participant
Masking Description: Group-I and Group-II will be blinded to the intervention while Group-III would not be administered an intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group-I (Control group) (Placebo Comparator): This group will be administered a placebo that is an odorless oil without any therapeutic effect)
  Interventions: Other: Placebo
- Group-II (Treated group) (Experimental): This group will be administered lavender oil.
  Interventions: Drug: Lavender Oil
- Group-III (Untreated group) (No Intervention): No intervention will be provided in this group.

INTERVENTIONS:
Drug: Lavender Oil — The oil used in this study will be lavender oil with a final concentration of 3% using almond oil (90%) as diluent. The oil after dilution and final preparation will be converted to proper clean vial in a fix amount (10 ml) and given to the students.
  Arms: Group-II (Treated group)
Other: Placebo — an odorless oil without any therapeutic effect
  Other Names: An odorless oil without any therapeutic effect
  Arms: Group-I (Control group)

SUMMARY:
Stress affects the health and is prevalent among medicine and pharmacy students. A number of factors such as busy schedules, course load and lack of recreational time during semesters as well as exams, have been reported to be associated with stress. Study reports that the use of aroma oils especially those with relaxant properties can alleviate the level of stress. This study aims to investigate the effects of aroma oils in stress during exams in pharmacy students.

DETAILED DESCRIPTION:
Stress is a disorder that affects human feelings through disturbance in behavior, thinking and mood. The mood disturbances further leads to mental, physical and emotional problems which affects the learning as well as thinking capabilities of individuals.Work load i.e. preparing for exams along with acquisition of knowledge, skills and attitudes have been reported as more stressful to cope up with, during university life of medical students. Exam load is reported as a major stressor and a number of studies have reported a suffering of 30% medical students due to exam stress. whereas some studies have reported a high stress level in 80% of college students during exams. No significant difference is observed for gender with regard to level of stress during exams. Besides course loads, exams, quizzes and busy schedule, academic competition among students for higher grades also promotes stress. This academic competition in students may sometimes be unavoidable. Alternative treatment namely aromatherapy, hydrotherapy and homeopathy are employed to reduce stress.

Aromatherapy is one of the alternative treatments in which oils extracted from natural sources such as flowers, petals and bark of plants are used to enhance the physical and psychological conditions of individuals. Various naturally extracted aromatic essences are applied in order to balance cognitive functions and memory retention. The aromatic essences/oils used in aromatherapy such as lavender oil, rosemary oil, jasmine oil, peppermint oil etc. are believed to stimulate cognitive function and are used for purposes of pain relieving, mood enhancement. Among these essences, lavender oil has been applied predominantly in oral administration, aromatherapy as well as massage therapy in many clinical studies exhibiting positive outcomes. Lavender oil reduces stress and produce relaxation via limbic system, particularly the amygdala and hippocampus.

A comparative study in 36 volunteers showed a reduced stress level in group using lavender oil as aromatherapy as compared to placebo group. Another study at Hong Kong University revealed the fact that aromatherapy may be utilized as an effective tool in order to alleviate pain, reduce depression and level of stress in older adults. A study in Iran among students, showed reduction in test-related anxiety with the use of Polianthes tuberosa essential oils. Similar study in students of Florida Atlantic University observed the vital effects of aroma oils and recommended the use of rosemary and lavender oil during exam for reducing stress level. In addition, lavender oil as stress reducer and leading towards relaxation during exam stress has been reported. Lavender oil as a cream along with a foot-bath, may be used in pregnant as well as non-pregnant females even, in order to reduce stress and anxiety. Based on aforementioned results, lavender oil may be effectively used to reduce the level of stress, produced due to any factor. However, none of the studies have reported the use of lavender oil in pharmacy students particularly during exams.

This study is aimed to target Pharmacy students at Imam Abdulrahman Bin Faisal University, Dammam, Saudi Arabia in order to evaluate the effect of aromatherapy i.e. lavender oil in stress among students during exams.

ELIGIBILITY:
Inclusion Criteria:

* The study includes only male student of Pharmacy college at IAU.
* Students from 2nd to 5th year are eligible for the study.
* All the students who are willing to participate voluntarily and are in healthy state will be included in the study.

Exclusion Criteria:

* Students from other colleges as well as female students are not included in the study.
* Any student who have no consent to participate will be excluded from this study.
* Students with a history of stress, anxiety and depression, with any serious chronic medical conditions, any known allergy to aromatherapy or lavender oil.

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study was conducted only in the male pharmacy students.
Enrollment: 49 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline perceived academic stress at day 7 and at day 14 | Day 1 to day 7 till day 14
  For investigating the level of stress during examination, a subjective perceived stress scale would be given to students to report perceived academic stress. The range of this scale is from 0 to 5 where a value of 0 indicate no academic stress and value of 5 indicate severe academic stress.
Change in baseline mean Blood pressure at day 7 and at day 14 | Day 1 to day 7 till day 14
  For observing any change in mean blood pressure, a blood pressure monitor will be used to determine any variation in blood pressure in millimeters of mercury (mm of Hg). A total of three readings will be taken at baseline day 0, day 7 and day 14. The mean value obtained from three readings will be considered final for each time point.
Change in baseline heart rate at day 7 and at day 14 | Day 1 to day 7 till day 14
  For observing any change in heart rate, a blood pressure monitor will be used to determine change in heart rate in beats per minute (BPM). A total of three readings will be taken at baseline, day 7 and day 14. The mean value obtained from three readings will be considered final for each time point.
Change in baseline Stool consistency at day 7 and day 14 | Day 1 to day 7 till day 14
  Bristol stool chart (BST) to indicate the consistency and frequency of stools passed during this period. Bristol stool chart consists of 7 types of stools. It is a subjective assessment.
Change in baseline headache at day 7 and day 14 | Day 1 to day 7 till day 14
  visual analog scale (VAS) for recording the intensity of headache experienced by students during this period. Visual Analogue Scale consist of a range of 1 to 5. (1 = normal and 5 = extreme). It is a subjective self reporting instrument.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Mastour S Al Ghamdi, PhD, Study Chair — Dean, College of Clinical Pharmacy
Locations (1):
- College of Clinical Pharmacy, Dammam, Eastern Province, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
All data pertaining to the clinical trial will be made available after study completion.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be available after March 5, 2018.